CLINICAL TRIAL: NCT05847894
Title: Assisting Pulmonary Disease Diagnosis With Ophthalmic Artificial Intelligence Technology
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen Third People's Hospital (Other); Guangzhou Kindness Health Care Center (Guangzhou Jiubang Shanxin Clinic Ltd), Guangzhou, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023KYPJ111
Record Dates: First submitted 2023-04-20; First posted 2023-05-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Diseases; Ophthalmological Diagnostic Techniques; Artificial Intelligence
Keywords: Pulmonary Diseases; Ophthalmological Diagnostic Techniques; Artificial intelligence
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: Individuals with one or more pulmonary diseases
  Interventions: Diagnostic Test: Ophthalmic examination; Diagnostic Test: Pulmonary Examination
- Control group: Individuals who do not suffer from pulmonary diseases
  Interventions: Diagnostic Test: Ophthalmic examination; Diagnostic Test: Pulmonary Examination

INTERVENTIONS:
Diagnostic Test: Ophthalmic examination — Various ophthalmic examination modalities, including slit lamp photography, fundus photography, optical coherence tomography imaging and optical coherence tomography angiography, etc.
Diagnostic Test: Pulmonary Examination — Various pulmonary examination modalities, including radiography, chest CT, pulmonary function measurement, etc.

SUMMARY:
This study intends to collect ophthalmologic examination results, pulmonary examination results and related indexes from patients with pulmonary disease and control populations, and combine big data analysis and artificial intelligence technology to explore whether new methods can be provided for early screening strategies for pulmonary disease with the aid of ophthalmologic examination, and thus assist in identifying the types of pulmonary disease and determining disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Those aged ≥18 years; or those aged <18 years who can cooperate with the relevant examination and are accompanied and informed by a guardian;
* People with respiratory-related diseases who were to undergo pulmonary examination, or those who volunteered to participate in the trial through publicity recruitment;
* expected survival time of 3 months or more;
* Those with no previous serious underlying disease and no history of serious eye disease;
* Those who can cooperate with ophthalmologic and pulmonary-related examinations and have regular follow-up examinations;
* Those who gave informed consent to the study prior to the trial and voluntarily signed the informed consent form;
* Other conditions that can be included in the study as judged by the investigator.

Exclusion Criteria:

* Patients who are unable to complete ophthalmology or pulmonary-related examinations and regular follow-ups due to serious diseases, trauma or surgery (serious ophthalmology diseases such as extremely poor vision that cannot be fixed, ocular atrophy, severe refractive interstitial clouding that prevents fundus photography, etc.);
* People with poor compliance due to various reasons such as alcohol or drug dependence, or mental disorders;
* Those without informed consent;
* Other conditions judged by the investigator to be unsuitable for participation in the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population was recruited from people who visited the cooperative medical unit for lung screening, and from people who were recruited through publicity at the unit and in the community.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic curve | Through study completion, an average of 1 year
  Determining the accuracy of diagnosing pulmonary disease with ophthalmic examination

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Kindness Health Care Center (Guangzhou Jiubang Shanxin Clinic Ltd), Guangzhou, Guangdong
  - the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Third People's Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided